CLINICAL TRIAL: NCT00638729
Title: Effects of Clonidine and Midazolam Premedication on Bispectral Index and Recovery After Elective Surgery
Brief Title: Clonidine Versus Midazolam for Premedication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Prof. Dr. J. Scholz, Chair of the Department of Anaesthesiology and Intensive Care Medicine, University Schleswig-Holstein Campus Kiel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A 157/01; A 157/01
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-02

CONDITIONS: Anxiety; Pain
Keywords: bispectral index; sedation; stress hormones; cognitive function
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Midazolam; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midazolam (Active Comparator): Pre-anesthetic medication with midazolam, 7.5 mg p.o., 60-90 min prior to estimated induction time
  Interventions: Drug: midazolam
- Clonidine (Active Comparator): pre-anesthetic medication with clonidine, 150 µg p.o., 60-90 min prior to estimated induction time
  Interventions: Drug: clonidine
- Placebo (Placebo Comparator): Pre-anesthetic medication with an inert tablet, p.o., 60-90 min prior to estimated induction time
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: midazolam — midazolam, 7.5 mg p.o., 60-90 min prior to estimated induction time
  Other Names: Dormicum
  Arms: Midazolam
Drug: clonidine — pre-anesthetic medication with clonidine, 150 µg p.o., 60-90 min prior to estimated induction time
  Other Names: Catapresan
  Arms: Clonidine
Drug: placebo — inert tablet p.o., 60-90 min prior to estimated induction time
  Arms: Placebo

SUMMARY:
alpha2-agonists like clonidine offer several useful effects that make these drugs an interesting alternative to benzodiazepines for pharmacological premedication. We therefore sought to determine the effect of pre-anesthetic medication with clonidine vs. midazolam in a randomized, double-blind, placebo controlled study. Effects of pre-anesthetic medication were assessed on (1) bispectral index (BIS),(2) sedation score and visual analog scales for anxiety and pain, (3) neuropsychologic tests to assess cognitive function and (4) circulating stress hormones.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* ASA physical status I and II
* informed consent
* weight 50 - 100 kg

Exclusion Criteria:

* cardiovascular disease
* pregnancy
* problems of consent due to mentally handicap or language.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Effect of premedication on bispectral index | prior study medication until 2 h postoperatively

SECONDARY OUTCOMES:
Effect of premedication on postoperative recovery | prior to study medication until 2 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, M.D., Study Chair — Chair of the Dept. of Anaesthesiology and Intensive Care Medicine, University of Schleswig-Holstein Campus Kiel
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University of Schleswig-Holstein Campus Kiel, Kiel, Germany

REFERENCES:
- [Background] Matot I, Sichel JY, Yofe V, Gozal Y. The effect of clonidine premedication on hemodynamic responses to microlaryngoscopy and rigid bronchoscopy. Anesth Analg. 2000 Oct;91(4):828-33. doi: 10.1097/00000539-200010000-00011. PMID 11004033
- [Background] Carabine UA, Milligan KR, Moore JA. Adrenergic modulation of preoperative anxiety: a comparison of temazepam, clonidine, and timolol. Anesth Analg. 1991 Nov;73(5):633-7. doi: 10.1213/00000539-199111000-00021. PMID 1683183
- [Background] Ghignone M, Quintin L, Duke PC, Kehler CH, Calvillo O. Effects of clonidine on narcotic requirements and hemodynamic response during induction of fentanyl anesthesia and endotracheal intubation. Anesthesiology. 1986 Jan;64(1):36-42. doi: 10.1097/00000542-198601000-00007. PMID 3942335
- [Background] Grottke O, Muller J, Dietrich PJ, Krause TH, Wappler F. [Comparison of premedication with clonidine and midazolam combined with TCI for orthopaedic shoulder surgery]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2003 Dec;38(12):772-80. doi: 10.1055/s-2003-45396. German. PMID 14666440
- [Background] Liu J, Singh H, White PF. Electroencephalogram bispectral analysis predicts the depth of midazolam-induced sedation. Anesthesiology. 1996 Jan;84(1):64-9. doi: 10.1097/00000542-199601000-00007. PMID 8572355
- [Background] Brosius KK, Bannister CF. Oral midazolam premedication in preadolescents and adolescents. Anesth Analg. 2002 Jan;94(1):31-6, table of contents. doi: 10.1097/00000539-200201000-00006. PMID 11772796
- [Background] Lindahl SG. The use of midazolam in premedication. Acta Anaesthesiol Scand Suppl. 1990;92:79-83; discussion 107. doi: 10.1111/j.1399-6576.1990.tb03191.x. PMID 2183537